CLINICAL TRIAL: NCT07017933
Title: Groundbreaking Renal Assist Device Intervening to ENhance cardioThoracic Surgery Outcomes
Acronym: GRADIENT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: 3ive Labs (Industry)
Collaborators: RQM+ (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GRADIENT 20-10
Record Dates: First submitted 2025-05-09; First posted 2025-06-12 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Renal Impairment After Cardiac Surgery; Renal Impairment; Acute Kidney Injury
Keywords: renal assist device; RAD; renal impairment; acute kidney disease; JuxtaFlow
MeSH Terms: conditions — Renal Insufficiency; Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Standard of Care (No Intervention): A standard bladder catheter (i.e. Foley) will be placed for bladder urine collection peri-operatively for up to 72 hours while in critical care. No JuxtaFlow catheters will be placed in control subjects.
- Renal Assist Device (Experimental): Subjects randomized to the Treatment group will receive up to 72 hours of controlled negative pressure (-15mmHg) into the renal pelvis of each kidney. Treatment will be discontinued when the subject is transferred out of critical care after at least 24 hours of treatment. A standard bladder catheter (i.e. Foley) will also be placed for bladder urine collection peri-operatively for up to 72 hours.
  Interventions: Device: Renal assist device

INTERVENTIONS:
Device: Renal assist device — The JuxtaFlow RAD includes two endoscopically placed ureteral catheters connected to a bedside pump system. The catheters are designed to deliver a mild, controlled negative pressure (-15 mmHg ± 2mmHg) into the renal pelvis of each kidney for up to 72 hours. This pressure is designed to diffuse through each of the million nephrons lowering intratubular pressure thereby improving the filtration gradient at the glomerulus while supporting overall kidney function.
  Other Names: RAD; JuxtaFlow
  Arms: Renal Assist Device

SUMMARY:
Patients with renal insufficiency who undergo cardiac surgery with cardiopulmonary bypass (CPB) are at significant risk for exacerbation of renal dysfunction postoperatively. This in turn is associated with an increased risk of prolonged intensive care unit (ICU) length of stay, other comorbidities including surgical complications and 30-day mortality. Renal impairment is generally identified based on an increase in serum creatinine concentration and/or a certain magnitude decrease in estimated glomerular filtration rate (eGFR).

The JuxtaFlow® Renal Assist Device (RAD) is designed to sustain or enhance glomerular filtration perioperatively for patients with renal insufficiency by applying a mild controlled negative pressure to the collecting system via the renal pelvis, thereby increasing effective filtration pressure and reducing tubular pressure. This mechanism is designed to support the kidneys' functions during times of renal stress that would be associated with intrarenal edema, volume overload, increased venous pressure, and inflammatory response. By supporting renal function, specifically during the acute stress of CPB, JuxtaFlow holds promise to protect nephron function, decrease renal hypoxia, and provide multifactorial kidney function support to maintain their ability to manage future stress.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for participation in this study, an individual must meet all the following criteria:

1. A candidate for elective or urgent on-pump coronary artery bypass grafting (CABG) and/or valvular surgery
2. Male or Female age 22 to 85 years
3. Estimated glomerular filtration rate (eGFR) 15 - 60 mL/min/1.73m2
4. Signed and dated informed consent
5. Female patients of childbearing potential must:

   1. have negative pregnancy test at the informed consent visit,
   2. be using previously initiated approved and effective contraception from the informed consent visit through completion of the study *The only recommended contraception is condoms.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Any individual, or their legally authorized representative (LAR), who does not understand the requests and risks of participating in the clinical trial or is unable to give informed consent
2. Pregnancy or lactation
3. Prior cardiac surgery within the last 6 months
4. Hemodynamic instability as determined by the Principal Investigator
5. Immunosuppression
6. Active infections (e.g. HIV, Tbc, and all types of Hepatitis)
7. History of polycystic kidney disease
8. Patients with only one active kidney or one poorly functioning kidney
9. Evidence of current kidney obstruction (e.g., Kidney stones)
10. Evidence of current hydronephrosis
11. Active upper and/or lower urinary tract infections
12. Malignancy; oncological Surgery within 5 years or ongoing antitumoral treatment
13. Ongoing sepsis or endocarditis
14. Patients who have an expected 30-day postoperative mortality greater than 10% as determined by the Principal Investigator
15. Any secondary condition as determined by the investigator that would place the subject at an increased risk or preclude the subject's full compliance with the study procedures, including injuries to the urinary organs and/or external genitals; or severe BPH
16. Unexplained/unexpected gross hematuria as determined by the Investigator
17. Current or planned treatment with an investigational drug (IND), device (IDE), or other investigational intervention within 3 months prior to or during participation in this clinical trial
18. Patients who have a current unrepaired ureteral avulsion as determined by the investigator
19. Patients otherwise contraindicated for urological interventions, including ureter guidewire placement via bladder cystoscopy and ureteral catheterization, or otherwise contraindicated for any of the other study procedures

Ages: 22 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2026-05-14 (Estimated); Study Completion 2026-06-14 (Estimated)

PRIMARY OUTCOMES:
Mean Peak Percent Change in Serum Creatinine | 96 hours peri-operative
  The mean peak percent change in serum creatinine from baseline values (prior to treatment) within the first 96 hours post-surgery for JuxtaFlow treated subjects as compared to controls.
Incidence of Treatment-Emergent Adverse Events | From enrollment to post-operative day 30
  The characterization and comparison of all types, frequency, and severity of adverse events (AEs) associated with JuxtaFlow treatment and controls.

SECONDARY OUTCOMES:
AUC Serum Creatinine | 96 hours peri-operative
  The area under the curve of serum creatinine changes from baseline values (prior to treatment) up to 96 hours post-surgery for JuxtaFlow treated subjects as compared to controls.
Creatinine Clearance | 24 to 48 hours post-operatively
  The average creatinine clearance as a measure of acute glomerular filtration rate, assessed for a minimum of 24 and up to 48 hours in 8-hour intervals during postoperative ICU JuxtaFlow treatment as compared to controls.
AKI incidence | From post-operative day 1 to 14
  The incidence of acute kidney injury (as determined by the KDIGO criteria) during post-surgical hospitalization and 14 days post-surgery with treatment as compared to controls.
Critical Care Length of Stay | through study study completion, an average of 1 year
  The post-surgical critical care length of stay (LOS) in the United States cohort for JuxtaFlow treated subjects as compared to controls.

OTHER OUTCOMES:
AKI severity | From post-operative day 1 to 14
  The severity and duration of acute kidney injury (as determined by the KDIGO criteria) during post-surgical hospitalization and 14 days post- surgery with treatment as compared to controls.
Urine Electrolytes | Up to 72 hours peri-operatively
  The change in urine sodium and potassium excretion rates during the treatment period (up to 72 hours) as compared to controls. Urine output will be assessed in 8-hour intervals perioperatively.
eGFR | From enrollment to post-operative day 30
  The change in eGFR (measured by 2021 EPI Cr method) measured at baseline, perioperatively, and at 14- and 30-days post-surgery in JuxtaFlow treated subjects as compared to controls.
Urine Output | Up to 72 hours peri-operatively
  The change in urine output (i.e. volume, urine flow, total oliguria time, total anuria time, etc.) over the course of treatment (up to 72 hours) as compared to controls. Urine output will be assessed in 8-hour intervals perioperatively.
Hospital Length of Stay | through study study completion, an average of 1 year
  The post-surgical hospital length of stay (LOS) in the United States cohort for JuxtaFlow treated subjects as compared to controls.
Anemia Incidence | through study study completion, an average of 1 year
  The incidence of anemia (as defined by a nadir hematocrit below 23% for women and 28% for men after initiating the investigational treatment) assessed immediately after starting treatment, immediately after surgery, and at every postoperative 8-hour period during treatment (up to 72-hours) after initiation of the treatment, and daily during the post-treatment period (until hospital discharge) as compared to controls.
Electrolyte abnormalities | through study study completion, an average of 1 year
  The incidence of electrolyte abnormalities (as defined by any alteration in the metabolic panel according to the reference values after initiating the investigational treatment) assessed immediately after starting JuxtaFlow treatment, immediately after surgery, and at every postoperative 8-hour period during treatment (up to 72-hours) after initiation of the investigational treatment, and daily during the post-treatment period (until hospital discharge). Assessed by comprehensive metabolic panel (includes calcium, sodium, potassium and carbon dioxide) and excretion rates calculated from a Urinalysis panel (includes sodium and potassium).
Azotemia | through study study completion, an average of 1 year
  The incidence of azotemia or elevated blood urea nitrogen (BUN).
Dialysis Incidence | From post-operative day 1 to 30
  The incidence of dialysis within 30 days post-surgery.
Hospital Readmission | From post-operative day 1 to 30
  Readmission to in-patient hospitalization for any reason within the 30- day postoperative period.
Mortality | From post-operative day 1 to 30
  All-cause mortality at 30 days post-surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Evelio Rodriguez, MD, Principal Investigator — Ascension Healthcare
Locations (1):
- Cleveland Clinic Florida, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rao VS, Maulion C, Asher JL, Ivey-Miranda JB, Cox ZL, Moreno-Villagomez J, Mahoney D, Turner JM, Wilson FP, Wilcox CS, Testani JM. Renal negative pressure treatment as a novel therapy for heart failure-induced renal dysfunction. Am J Physiol Regul Integr Comp Physiol. 2021 Oct 1;321(4):R588-R594. doi: 10.1152/ajpregu.00115.2021. Epub 2021 Aug 18. PMID 34405731
- See also: Roivios Studies — https://roivios.com/studies/